CLINICAL TRIAL: NCT00654641
Title: Prevention of Abdominal Wound Complications After Cesarean Delivery in Obese Women Utilizing Negative Pressure Wound Therapy
Brief Title: Prevention of Wound Complications After Cesarean Delivery in Obese Women Utilizing Negative Pressure Wound Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment. No apparent treatment effect.
Sponsor: West Virginia University (Other)
Collaborators: CAMC Health System (Other)
Responsible Party: Principal Investigator, Michael Stitely, Adjunct Associate Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-20292
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2012-12

CONDITIONS: Surgical Wound Dehiscence; Wound Infection
Keywords: Surgical Wound Dehiscence; Wound Infection; Obesity; Cesarean Delivery; Wound Closure; Negative Pressure wound closure
MeSH Terms: conditions — Surgical Wound Dehiscence; Wound Infection; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Negative pressure wound closure (Experimental): Negative Pressure wound closure
  Interventions: Procedure: Negative pressure wound closure
- Standard wound closure (Active Comparator): Standard Wound Closure
  Interventions: Procedure: Standard wound closure

INTERVENTIONS:
Procedure: Negative pressure wound closure — Applying negative pressure to primary wound closure
  Arms: Negative pressure wound closure
Procedure: Standard wound closure — Standard wound closure
  Arms: Standard wound closure

SUMMARY:
Wound complications after Cesarean section (C-section) are common in obese women. Approximately 25% of obese women having a C-section will have a wound complication. This research study is designed to assess whether applying a source of vacuum (suction) to the wound can reduce the risk of wound complications. The investigators plan to enroll 220 women into the study.

Women will be randomly selected to receive standard stitching and stapling of the incision (cut on the abdomen) or closure with stitches, staples and wound suction. Subjects will be seen for follow-up visits in 7-14 days and again at 4-6 weeks after surgery. The number of wound complications in each group will be compared. If the wound suction technique is successful in preventing wound complications, this may substantially reduce pain and suffering in a large number of women undergoing C-section for delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing Cesarean delivery.
2. Patient at least 18 years of age.
3. Weight greater than 199 pounds.
4. Depth of subcutaneous tissue (measured from fascia to epidermis) of greater than or equal to 4 centimeters.

Exclusion Criteria:

1. Weight less or equal to 199 pounds or less than 4 cm of subcutaneous tissue present.
2. Inability to give proper informed consent.
3. Inability to adhere to follow-up provisions of the study (return for 2 post-operative visits at 7-14 days post-op and between 4-6 weeks post-op).
4. Patient less than 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Stitely, MD, Principal Investigator — West Virginia University
Locations (2):
- United States (2):
  - CAMC Women and Children's Hospital, Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Pressure Wound Closure: Negative Pressure wound closure utilizing wall suction and a drain placed exterior to the closed wound.
- Standard Wound Closure: Wound closed in standard fashion utilizing subcutaneous absorb-able suture and skin staples.
Period: Overall Study
Arm/Group | Negative Pressure Wound Closure | Standard Wound Closure
Started | 28 | 26
Completed | 26 | 23
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Closure | Standard Wound Closure | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Patients Experiencing a Wound Complication
Description: Superficial or deep space surgical site infection, or any type of wound disruption, including wound hematoma or seroma.
Time Frame: 6 Weeks post-partum
Measure: Number; unit: Participants
Arm/Group | Negative Pressure Wound Closure | Standard Wound Closure
Number analyzed (Participants) | 28 | 26
Participants | 15 | 10

ADVERSE EVENTS:
Arm/Group | Negative Pressure Wound Closure | Standard Wound Closure
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 15/28 | 10/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Pressure Wound Closure (N=28) | Standard Wound Closure (N=26)
Wound complication (Skin and subcutaneous tissue disorders) | 15 (15) | 10 (10) — Any wound complication including superficial or deep surgical site infection, wound disruption, hematoma or seroma.

LIMITATIONS AND CAVEATS:
Slow enrollment caused the closure of the trial prior to meeting enrollment target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No